CLINICAL TRIAL: NCT04002167
Title: A Novel Neuromonitoring Guided Cognitive Intervention for Targeted Enhancement of Working Memory
Brief Title: A Novel fNIRS Neurofeedback Intervention for Enhancement of Working Memory in Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Hadi Hosseini, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 328066; R61MH119289 (NIH)
Record Dates: First submitted 2019-06-24; First posted 2019-06-28 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: ADHD
Keywords: ADHD; Working memory; functional near infrared spectroscopy (fNIRS); magnetic resonance imaging (MRI); Neurofeedback; Cognitive training; Neuromonitoring
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Neurofeedback; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neurofeedback (Experimental): The Neurofeedback group will receive 12 sessions of computerized cognitive intervention combined with neurofeedback in the lab.
  Interventions: Behavioral: Neurofeedback
- Cognitive Training (Active Comparator): The Cognitive Training group will receive 12 sessions of computerized cognitive intervention in the lab.
  Interventions: Behavioral: Cognitive training
- Waitlist (No Intervention): Both Neurofeedback and Cognitive Training groups will be assigned to waitlist before starting the corresponding intervention.

INTERVENTIONS:
Behavioral: Neurofeedback — The Neurofeedback group will receive the proposed intervention which integrates computerized working memory training with neuromonitoring and neurofeedback.
  Arms: Neurofeedback
Behavioral: Cognitive training — The Cognitive training group will receive computerized working memory training with performance feedback.
  Arms: Cognitive Training

SUMMARY:
The proposed study is to test and validate a novel intervention that integrates computerized cognitive training with real-time neuromonitoring and neurofeedback to enhance working memory by probing the individualized neural systems underlying working memory. We will test the proposed intervention on children with ADHD with working memory deficits. The R61 proof-of-concept phase will assess the target engagement, effective dose and feasibility.

ELIGIBILITY:
Inclusion criteria include:

* Age from 7 to 11 years
* Diagnosis and/or current symptoms of ADHD
* Full-scale Intelligence quotient (IQ) ≥80
* Behavior Rating Inventory of Executive Functions (BRIEF), Working Memory Scale t-score > 65
* Allowed comorbidities include oppositional defiant disorder, learning disabilities excluding dyslexia, and mild anxiety and/or depression.

Exclusion criteria:

* Presence of severe neurological or psychiatric disease other than those allowed under inclusion
* Sensory deficits that would preclude participation in assessments or imaging
* History of significant head trauma with loss of consciousness
* Contraindications to MRI (e.g. metal implants or claustrophobia)
* Enrollment in other intervention studies

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hadi Hosseini, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Neurofeedback (Phase I): The Neurofeedback group will receive 12 sessions of computerized cognitive intervention combined with neurofeedback in the lab.
- Waitlist (Phase I): Both Neurofeedback and Cognitive Training groups will be assigned to waitlist before starting the corresponding intervention.
- Cognitive Training (Phase II): The Cognitive Training group will receive 12 sessions of computerized cognitive intervention in the lab.
Period: Overall Study
Arm/Group | Neurofeedback (Phase I) | Waitlist (Phase I) | Cognitive Training (Phase II)
Started | 33 | 32 | 0
Completed | 21 | 15 | 0
Not Completed | 12 | 17 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol are included in the analyses
Groups:
- Total: Total of all reporting groups
Arm/Group | Neurofeedback (Phase I) | Waitlist (Phase I) | Total
Number analyzed (Participants) | 21 | 15 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 15 | 36
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 12 | 8 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 10 | 18
  More than one race | 9 | 3 | 12
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 15 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Target Frontal-parietal Activity
Description: Change in activity in the target frontal-parietal network measured by functional near infrared spectroscopy (fNIRS) during an N-back working memory task. A general linear model is applied to recorded signal and the beta coefficients from the model are extracted as a proxy for brain activity in fronto-pariteal network which subserves working memory function. There is no established population mean for beta coefficient of brain activity. Higher (lower) beta coefficients reflect higher (lower) activation in the target brain network. A positive change indicates increased brain activity. Increased frontal-parietal activity reflects better engagement of this brain network during working memory performance.
Time Frame: baseline and 6 weeks
Population: Participants with usable data are included in the analysis
Measure: Mean (Standard Deviation); unit: beta coefficient
Arm/Group | Neurofeedback (Phase I) | Waitlist (Phase I)
Number analyzed (Participants) | 20 | 14
beta coefficient | 2.31 (1.73) | -4.74 (2.50)

2. Primary Outcome: Change in Working Memory Performance
Description: Accuracy in an N-back working memory task was calculated as the percentage of correct responses to target stimuli.
Time Frame: baseline and 6 weeks
Population: Participants with usable data are included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change in accuracy
Arm/Group | Neurofeedback (Phase I) | Waitlist (Phase I)
Number analyzed (Participants) | 20 | 14
percent change in accuracy | 2.12 (15.70) | -0.53 (12.09)

3. Secondary Outcome: Change in Behavior Rating Inventory of Executive Function (BRIEF), Working Memory T-score
Description: BRIEF assesses everyday behavior associated with specific domains of the executive functions. BRIEF working memory T-score ranges from <30 to >100 with higher scores indicating larger impairment in working memory. Lower T-scores on BRIEF indicates better working memory. T-score of 50 indicates the population mean with a standard deviation of 10. BRIEF working memory T-score of 65 and higher is indicative of deficits in working memory.
Time Frame: baseline and 6 weeks
Population: Participants with usable data are included in the analysis.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Neurofeedback (Phase I) | Waitlist (Phase I)
Number analyzed (Participants) | 21 | 15
t-score | -8.4 (6.1) | -0.85 (7.94)

4. Secondary Outcome: Change in Wide Range Assessment of Memory and Learning 2 (WRAML-2), General Memory Index Score
Description: WRAML-2 assesses clinical issues in learning and memory functions. WRAML-2 Working Memory Index score ranges from 50 to 150 with higher scores indicating better working memory performance
Time Frame: baseline and 6 weeks
Population: Participants with usable data were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neurofeedback (Phase I) | Waitlist (Phase I)
Number analyzed (Participants) | 18 | 14
score on a scale | 6.6 (16.36) | 9.38 (11.21)

5. Secondary Outcome: Change in Conners 3rd Edition ADHD Index Score
Description: Conners 3 will be used to measure changes in clinical ADHD symptoms. Conners 3 ADHD index score ranges from 0 to 100 with higher scores indicating elevated ADHD symptoms. Conners 3 ADHD index score of higher than 65 is indicative of ADHD diagnosis.
Time Frame: baseline and 6 weeks
Population: Participants with usable data were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neurofeedback (Phase I) | Waitlist (Phase I)
Number analyzed (Participants) | 21 | 15
score on a scale | -6.21 (10.61) | -1 (3.49)

6. Secondary Outcome: Change in Conners 3rd Edition Inattention T-score
Description: Conners 3 will be used to measure changes in clinical inattention symptoms. Conners 3 inattention t-score ranges from <30 to >100 with higher scores indicating larger impairment in attention. T-score of 50 indicates the population mean with a standard deviation of 10. Inattention t-score of 65 and higher is indicative of deficits in attention.
Time Frame: baseline and 6 weeks
Population: Participants with usable data were included in the analysis.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Neurofeedback (Phase I) | Waitlist (Phase I)
Number analyzed (Participants) | 21 | 15
t-score | -4.8 (11.3) | 0.41 (6.38)

7. Secondary Outcome: Change in Developmental NEuroPSYchological Assessment II (NEPSY-II) Composite Score
Description: NEPSY-II consists of a set of subtests measuring cognitive functions required for success in school. The subtests include auditory attention & response, inhibition, word-list interference, and comprehension of instructions. The composite scores were quantified by averaging the scores across sub-scales. A positive change in composite score suggests increased ability in subtest domains. The composite score below 8 suggest deficits. The composite scores range from 0 to 20; lower scores correspond to more deficits, and higher scores correspond to more abilities.
Time Frame: baseline and 6 weeks
Population: participants with usable data were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neurofeedback (Phase I) | Waitlist (Phase I)
Number analyzed (Participants) | 21 | 15
units on a scale | 0.72 (2.56) | 1.05 (2.79)

8. Other Pre Specified Outcome: Change in Continuous Performance Test (CPT) Accuracy
Description: CPT is standard test for measuring vigilance, sustained attention and inhibitory control.
Time Frame: baseline and 6 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in California Verbal Learning Test - Children's Version (CVLT-C) Score
Description: CVLT-C test measures performance in learning and recalling verbal materials
Time Frame: baseline and 6 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Parent Stress Index 4th Edition (PSI-IV)
Description: PSI-IV evaluates the magnitude of stress in the parent-child system
Time Frame: baseline and 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 months
Arm/Group | Neurofeedback (Phase I) | Waitlist (Phase I)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 1/33 | 0/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neurofeedback (Phase I) (N=33) | Waitlist (Phase I) (N=32)
feeling of heat in an eye (Eye disorders) | 1 | 0 — Unrelated to treatment

LIMITATIONS AND CAVEATS:
The study did not achieve the planned number of participants with usable data due to halt in the study due to COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT04002167/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT04002167/SAP_001.pdf